CLINICAL TRIAL: NCT03294161
Title: Transition-state Analog Inhibitor of Human Purine Nucleoside Phosphorylase as an Adjunct in Cutaneous Leishmaniasis Therapy: a Randomized and Controlled Trial
Brief Title: Fourth-generation Immucillin Derivative DI4G Associated Therapy in Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Federal University of Bahia (Other); Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Fernanda V Prates, MD, MSc, Principal Investigator, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Immucillin DI4GTrial
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Leishmaniasis; Leishmaniasis, Cutaneous; Leishmaniasis; American
Keywords: Meglumine antimoniate; L.Braziliensis; Immunotherapy; Immucillin
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Cutaneous; Leishmaniasis, Mucocutaneous | interventions — Meglumine Antimoniate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immucillin DI4G (Experimental): Meglumine Antimoniate by intravenous route at 20mg/kg/day during 20 days + Immucillin DI4G 2% by topical use once a day at the ulcer for 20 days .
  Interventions: Drug: Immucillin DI4G
- Meglumine Antimoniate (Active Comparator): Meglumine Antimoniate by intravenous route at 20mg/kg/day during 20 days + placebo for topical use once a day at the ulcer for 20 days.
  Interventions: Drug: Meglumine antimoniate

INTERVENTIONS:
Drug: Immucillin DI4G — Immucillin DI4G was administered by topical use at 2% concentration once a day for 20 days associated with Meglumine antimoniate administered by intravenous route at a dosage of 20mg/kg/day, during 20 days.
  Other Names: Fourth-generation Immucillin Derivative
  Arms: Immucillin DI4G
Drug: Meglumine antimoniate — Placebo for topical use once a day at the ulcer for 20 days associated with Meglumine antimoniate administered as the standard treatment for cutaneous leishmaniasis by intravenous route at a dosage of 20mg/kg/day, during 20 days.
  Other Names: Glucantime
  Arms: Meglumine Antimoniate

SUMMARY:
A clinical trial to asses efficacy and safety of Transition-state Analog Inhibitor of Human Purine Nucleoside Phosphorylase for topical use associated standard antimonial in the treatment of Cutaneous Leishmaniasis in Bahia, Brazil.

DETAILED DESCRIPTION:
The treatment of cutaneous leishmaniasis caused by L. braziliensis in Brazil with pentavalent antimony is associated with a high rate of failure, reaching up to 45% of cases. Additionally, pentavalent antimony is only administered by parenteral route with important toxicity and ulcer lesion healing takes a long time, from 2 to 3 months.

So, this randomized and controlled clinical trial was designed to compare the efficacy and safety of standard antimonial (20mg/day /kg for 20 days) associated with Transition-state Analog Inhibitor of Human Purine Nucleoside Phosphorylase for topical use versus standard antimonial (20mg/kg/day for 20 days) associated with placebo for topical use in the treatment of Cutaneous Leishmaniasis and Early Cutaneous Leishmaniasis caused by L. braziliensis in the endemic area of Corte de Pedra, Bahia, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (untreated) cutaneous leishmaniasis or early cutaneous leishmaniasis with localized lesions and a positive culture or diagnosed by polymerase chain reaction (PCR) methods or by intradermal skin testing (Montenegro test).
* Number of lesions: 1 to 3 ulcerative lesions.
* Lesion´s diameter: 1 to 5 cm.
* Disease duration: up to three months.

Exclusion Criteria:

* Aspartate aminotransferase, alanine aminotransferase >3 times upper limit of normal range
* Serum creatinine or blood urea nitrogen >1.5 times upper limit of normal range
* Evidence of serious underlying disease (cardiac, renal, hepatic or pulmonary)
* Immunodeficiency or antibody to HIV
* Any non-compensated or uncontrolled condition, such as active tuberculosis, malignant disease, severe malaria, HIV, or other major infectious diseases
* Lactation, pregnancy (to be determined by adequate test) or inadequate contraception in females of childbearing potential for treatment period plus 2 months
* Negative parasitology (aspirate/biopsy/PCR) or negative Montenegro test
* Any history of prior anti-leishmania therapy
* Any condition which compromises ability to comply with the study procedures
* Lack of ability or willingness to give informed consent (patient and/or parent / legal representative)
* Anticipated non-availability for study visits/procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Cure rate or complete cicatrization of the ulcer. | 6 months after treatment
  Bidirectional measurements of ulcers will be taken of the patients' lesions at the initial visit, and at each follow-up visit with standardized caliper. The area involved will be calculated as the product of the two measurements.
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients.

SECONDARY OUTCOMES:
Initial cure rate or complete cicatrization of the ulcer. | 2 months after treatment
  Bidirectional measurements of ulcers will be taken of the patients' lesions at the initial visit, and at each follow-up visit with standardized caliper. The area involved will be calculated as the product of the two measurements.
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Edgar M Carvalho, MD, PhD, Principal Investigator — Federal University of Bahia; Paulo RL Machado, MD, PhD, Study Chair — Federal University of Bahia
Locations (1):
- Corte de Pedra Health Post, Corte de Pedra, Estado de Bahia, Brazil